CLINICAL TRIAL: NCT04650919
Title: Placement of a Laryngeal Allograft Aortic Implant After Total Laryngectomy to Rehabilitate Laryngeal Function
Brief Title: Aortic Laryngeal Rehabilitation Graft
Acronym: GRAAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7649
Record Dates: First submitted 2020-11-16; First posted 2020-12-03 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Laryngeal Cancer; Total Laryngectomy
Keywords: laryngectomy
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Procedure: Total laryngectomy and reconstruction by stented aortic allograft (using human tissue and device).

INTERVENTIONS:
Procedure: Total laryngectomy and reconstruction by stented aortic allograft (using human tissue and device). — The procedure consists of 2 operating times:
  * Surgery S1 (1st surgical procedure): total laryngectomy and placement of the stented aortic graft (human tissue + device: NOVATECH GSS TM (trademark) TD), under tracheotomy cover.
  * Surgery S2 (2nd surgical procedure) (between S1 +24 weeks and S1 +36 weeks) : opening of the proximal part of the graft by endoscopic way with maintenance of the tracheotomy orifice to ensure patient safety.

SUMMARY:
The larynx is a cartilaginous organ of the respiratory system located in the throat, which plays an essential role in respiratory function, swallowing and sound production.

In the case of advanced tumours, the surgical option most often remains total laryngectomy, with the corollary of a major impact on quality of life, not so much because of the loss of voice, but because of the presence of a definitive tracheostoma with particularly deleterious consequences.

The majority of the work of the different teams around the world has focused on restoring phonatory function, but no technique - apart from the artificial larynx developed in the ENT department of the Hautepierre Hospital - has yet succeeded in removing the tracheotomy orifice, requiring the restoration of a common passage between the respiratory and swallowing passages. If nutrition and phonatory function can still be supplemented after such an operation (oesophageal rehabilitation, implant placed between the trachea and oesophagus), natural breathing is no longer possible. Patients are forced to wear a permanent tracheotomy opening.

There are currently only 2 ways to try to restore all the functions of the larynx after total laryngectomy: i) laryngeal transplantation, but this procedure requires maintaining immunosuppressive treatment, which is not possible in patients suffering from cancer of the larynx, which is not a vital organ, ii) artificial larynx made of biomaterials (titanium), the first cases of which were performed worldwide in the ENT department of the Strasbourg University Hospital in 2012, results published in the NEJM (API 2008-2009 HUS No. 4493- IDRCB No.: 2011-A00032-39. However, difficulties were encountered with the use of the titanium prosthesis due to the bulk and rigidity of the removable and non-removable part, which caused residual swallowing difficulties (false routes).

It is now possible, due to the development of new allograft techniques in humans for tracheal replacement (studies published on a large number of cases with several years of hindsight, cf. references), to switch to the "all biological" using an aortic graft stented with a silicone stent. We wish to use these grafts in laryngeal restoration after total laryngectomy by our team, while exploiting all the data and experience acquired (unique in the world) within the ENT department of Hautepierre Hospital. This new conceptual leap should make it possible to significantly improve the patient's quality of life and the performance previously acquired in clinical trials on the artificial larynx in its entirety (breathing, phonation) or partially (swallowing).

The investigators thus propose to evaluate this new artificial larynx in aortic allograft, the objective of which is to supplement the respiratory, swallowing and phonation functions in patients laryngectomized for carcinological causes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with carcinomatous pathology of the upper airways requiring total laryngectomy
* Patient affiliated to a social health insurance scheme (beneficiary or beneficiary's successor)
* Patient speaks and reads French, understands the objectives and risks of the research and is able to provide dated and signed informed consent.
* Patient having been informed of the results of the prior medical examination
* For a woman with the ability to procreate: negative blood pregnancy test (verified during preoperative blood work) and effective contraception throughout the study.

Exclusion Criteria:

* Patient with a contraindication to general anaesthesia and/or iodinated contrast agents
* Breastfeeding woman
* Patient with a WHO performance index of grade strictly greater than 2 at the inclusion visit
* Patient with subglottic or basi-lingual tumour extension greater than 1 cm (by endoscopic control and CT scan)
* Patient having undergone cervico-facial radiotherapy prior to surgical management
* Patient suffering from severe coagulation disorders (checked during the blood test performed as part of the standard care to make the diagnosis of cancer)
* Patient with a history of allergy to DMSO, DHEA, clindamycin, gentamicin, vancomycin used for graft treatment and preservation
* Inability to give informed information about the patient (patient in emergency situations, difficulties in understanding the patient)
* Patient in exclusion period (determined by a previous or ongoing study)
* Patient under safeguard of justice
* Patient under guardianship,curatorship, family guardianship
* Any situation considered by the operating physician as falling under a non-inclusion criterion
* Patient suffering from a decompensated psychiatric pathology or at risk of decompensation, which may interfere with the follow-up modalities in the research setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Success or Failure of the procedure | 6 month following the second surgery (Month 6; Visit 6)
  The primary endpoint is composite, combining clinically assessments:
  * the score on the Respiratory Function Assessment (clinically assessed : 0: no dyspnea, to 3 (major dyspnea) and
  * the score (0-3) on the Swallowing Ability Assessment (0: no issue to 3: major food misdirection) assessed by nasofibroscopy.
  The procedure will be considered a success if :
  * respiratory function: no dyspnea (score=0) or moderate dyspnea (score=1) AND
  * swallowing ability: no false-route (score=0) or moderate false-route (score=1)
  In all other cases, the procedure will be considered a failure.

SECONDARY OUTCOMES:
Scoring of dyspnea at each follow-up visit | 1 to 8 days and15 days following the second surgery (Visit 3), Month 1 (Visit 4), Month 3 (Visit 5), Month 6 (Visit 6), Month 9 (Visit 7) and Month 12 (Visit 8)
  Score on the Respiratory Function Assessment (clinically assessed : 0: no dyspnea, to 3 (major dyspnea)
Scoring of swallowing ability assessment at each follow-up visit | 8 days and 15 days following the second surgery (Visit 3), Month 1 (Visit 4), Month 3 (Visit 5), Month 6 (Visit 6), Month 9 (Visit 7) and Month 12 (Visit 8)
  Score (0-3) on the Swallowing Ability Assessment (0: no issue to 3: major food misdirection) assessed by nasofibroscopy.
Evaluation of the patient's voice by the "Voice Handicap Index 30" (Pommée, 2018) | 8 days and 15 days following the second surgery (Visit 3), Month 1 (Visit 4), Month 3 (Visit 5), Month 6 (Visit 6), Month 9 (Visit 7) and Month 12 (Visit 8)
  The Voice Handicap Index is a scale where the patient grades the severity of his disorder by 10 items on a scale from 0 (never) to 4 (always). Close to 0 may consider that the disability is almost nil, close to 120 the patient's voice has a significant impact on his or her daily life.
Analysis of Adverse Events and Serious adverse Events throughout the study | From the signature of the consent form (inclusion visit) to the end of study visit, up to 28 months.

CONTACTS AND LOCATIONS:
Overall Officials: Christian DEBRY, MD PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- ENT department-Hôpitaux Universitaires de Strasbourg, Strasbourg, France